CLINICAL TRIAL: NCT00167414
Title: A Phase II Study for Using Radiosurgery on Limited Metastases of Breast Cancer
Brief Title: Study for Using Radiosurgery on Limited Metastases of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hong Zhang, Assistant Professor Department of Radiation Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 8700
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer, Metastatic
Keywords: conformal radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypofractionated Stereotactic Body Radiation Therapy (Experimental): Use of Hypofractionated Stereotactic Body Radiation Therapy for limited metastases with breast cancer primary.
  Interventions: Procedure: Hypofractionated Stereotactic Body Radiation Therapy; Radiation: Hypofractionated Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Hypofractionated Stereotactic Body Radiation Therapy — Hypofractionated Stereotactic Body Radiation Therapy
Radiation: Hypofractionated Stereotactic Body Radiation Therapy — Hypofractionated Stereotactic Body Radiation Therapy for treatment of limited metastases from breast cancer primary.

SUMMARY:
The purpose of this study is to evaluate whether radiosurgery, along with standard chemotherapy, immunotherapy (the treatment of cancer by modulating the immune system and immune response), or hormonal therapy, affects the quality and length of life. The standard therapy is surgery, radiation therapy, or chemotherapy alone or in any combination. A second purpose of this study is to determine if the levels of a special type of protein (called cytokines) found in the blood are related to the quality of life while on this treatment.

DETAILED DESCRIPTION:
Before treatment begins, you will have a physical exam and blood tests. Physical evaluations and blood tests will be done each week while you are receiving treatment, and at follow-up visits. You will be seen for follow-up evaluations 4 weeks after treatment is completed, and every three months thereafter. You will be asked to fill out a Quality of Life questionnaire, which should take 5-10 minutes to complete. This will be done prior to treatment and at your follow-up visits. You will receive high dose radiation therapy directed at the site of metastasis. This treatment will be given once a day, 5 times a week (Monday through Friday) for one to four weeks depending on the location and size of the disease to be treated.

ELIGIBILITY:
Inclusion Criteria:

* Age: no limit
* Karnofsky performance status (KPS) ≥ 70
* No more than 5 metastatic sites involving one or more different organs (liver, lung or bone).
* The size of the lesion must be such that it can be safely treated to sterilizing radiation doses according to the rules in the protocol.
* Previously treated lesions are not eligible unless the prescribed dose can be safely delivered.
* Concurrent therapy is allowed and recommended. The chemotherapy protocol type and schedule are at the discretion of the medical oncologist.
* Informed consent must be obtained.
* Pregnancy test must be negative for women of child bearing potential

Exclusion Criteria:

* Inability of patient to be followed longitudinally as specified by protocol.
* Technical inability to achieve required dose based on safe dose constraints required for radiosurgery.
* Women who are pregnant or nursing.
* Failure to meet requirements in Inclusion Criteria
* Contraindications to radiation.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-12 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, MD, Principal Investigator — University of Rochester
Locations (1):
- Department of Radiation Oncology: University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Using Radiosurgery On Limited Metastases Of Breast Cancer — http://radonc.urmc.rochester.edu/novalis_brochure/breast_mets_study.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Started | 49
Completed | 39
Not Completed | 10
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The percent of patients that survived from date of enrollment until 2 year follow-up visit.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
percentage of participants | 74

2. Primary Outcome: Overall Survival
Description: The percent of patients that survived from date of enrollment until 4 year follow-up visit
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
percentage of participants | 54

3. Primary Outcome: Overall Survival
Description: The percent of patients that survived from date of enrollment until 6 year follow-up visit
Time Frame: 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
percentage of participants | 47

4. Secondary Outcome: Percent of Patients With Lesion Local Control
Description: Lesion local failure was scored as an event if any treated lesion increased by greater than or equal to 20% using the Response Evaluation Criteria in Solid Tumors criteria or local failure was confirmed pathologically. Lesion control includes all participants that did not fall into the category of lesion failure.
Time Frame: 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
percentage of participants | 87

5. Secondary Outcome: Number of Participants Who Experienced a Grade 4 or 5 Toxicity
Description: Number of participants who experienced a grade 4 or 5 toxicity
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 39
Participants | 0

ADVERSE EVENTS:
Arm/Group | Hypofractionated Stereotactic Body Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Stereotactic Body Radiation Therapy (N=39)
nonmalignant pleural and pericardial effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes